CLINICAL TRIAL: NCT06923280
Title: Efficacy and Safety of Pegylated Interferon Therapy in Chronic Hepatitis B Patients After Discontinuation of Antisense Oligonucleotide or Small Interfering RNA: A Prospective, Adaptive, Open-label, Randomized Controlled Study
Brief Title: Sequential PEG-IFN for HBV After Ending RNA-targeted Regimens
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Huashan Hospital (Other)
Responsible Party: Principal Investigator, Wen-hong Zhang, Director of Division of Infectious Diseases, Huashan Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SPHERE
Record Dates: First submitted 2025-04-03; First posted 2025-04-11 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Hepatitis B, Chronic
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- A：Immediate PEG-IFNα Induction (Experimental): Receive PEG-IFNα for 24 weeks, followed by 24-week treatment-free follow-up
  Interventions: Drug: Pegylated Interferon-alpha (IFN)
- B: Deferred PEG-IFNα Initiation (Experimental): Undergo 24-week observation, then receive PEG-IFNα for 24 weeks
  Interventions: Drug: Pegylated Interferon-alpha (IFN)

INTERVENTIONS:
Drug: Pegylated Interferon-alpha (IFN) — pegylated interferon-alpha 180 μg once weekly for 24 weeks

SUMMARY:
The goal of this clinical trial is to compare sequential PEG-IFNα therapy strategies in chronic hepatitis B (CHB) patients previously treated with ASO/siRNA. The main questions it aims to answer are:

1. Does sequential PEG-IFNα therapy (vs. deferred/no treatment) improve HBsAg clearance rates?
2. What are the HBsAg clearance and relapse rates after 24 weeks of PEG-IFNα therapy?
3. Is intermittent PEG-IFNα therapy as effective and safe as continuous therapy?

Researchers will compare:

• Group A (immediate 24-week PEG-IFNα + 24-week follow-up) vs. Group B (24-week observation + 24-week PEG-IFNα) in Phase 1 to see if sequential PEG-IFNα therapy will improve HBsAg loss rate .

Researchers will describe:

* The response rate of IFN treatment in non-responders (HBsAg-positive) in Phase 2.
* The relaspe rate of responders (HBsAg-negative).

Participants will:

Phase 1 (0-48 weeks):

* Group A: Receive PEG-IFNα for 24 weeks, followed by 24-week treatment-free follow-up.
* Group B: Undergo 24-week observation, then receive PEG-IFNα for 24 weeks.

Phase 2 (48-96 weeks):

* HBsAg-positive at week 48 patients either from group A or group B : Receive 24-week PEG-IFNα therapy, followed by 24-week follow-up.
* HBsAg-negative at week 48 patients either from group A or group B: Enter 24-week follow-up without treatment.

All participants will undergo:

• HBsAg quantification, HBV DNA, liver function, and safety monitoring (every 12 weeks).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years.
* Chronic HBV infection (documented HBsAg positivity for >6 months).
* Prior participation in ASO or siRNA clinical trials:
* Received ≥1 dose of ASO/siRNA (or matched placebo, if applicable).
* Achieved ≥1 log10 IU/mL HBsAg decline from baseline during prior therapy.
* Discontinued ASO/siRNA therapy before screening.
* Screening HBsAg: 0.05-500 IU/mL.
* No prior interferon (IFN) therapy within 6 months before enrollment.
* Willingness to comply with study-related treatments, tests, and procedures.
* Commitment to contraception during the study.
* Voluntary participation with signed informed consent.

Exclusion Criteria:

* Decompensated cirrhosis or hepatic malignancy (evidenced by imaging or histology within 6 months before/during screening).
* Elevated AFP: Screening AFP >100 ng/mL; AFP 20-100 ng/mL with imaging-confirmed hepatocellular carcinoma (ultrasound/CT/MRI).
* Coinfection with hepatitis A virus (HAV), hepatitis C virus (HCV), hepatitis D virus (HDV), hepatitis E virus (HEV), or human immunodeficiency virus (HIV).
* Recent immunomodulatory therapy: Systemic corticosteroids, thymosin, or other potent immunomodulators for >2 weeks within 6 months before enrollment.
* Pregnancy, lactation, or plans for pregnancy during the study.
* Autoimmune hepatitis.
* Active autoimmune diseases (e.g., psoriasis, systemic lupus erythematosus).
* Uncontrolled cardiovascular disease (e.g., unstable angina, myocardial infarction within 6 months).
* Poorly controlled endocrine disorders (e.g., diabetes mellitus, thyroid dysfunction).
* Severe psychiatric disorders: History of depression, anxiety, bipolar disorder, schizophrenia, or family history of psychiatric conditions (especially depression).
* Substance abuse: Alcohol (>40 g/day for males; >20 g/day for females) or Illicit drug use.
* Severe retinopathy or ophthalmologic disorders.
* Renal diseases: Chronic nephritis, renal insufficiency, nephrotic syndrome.
* Major organ dysfunction (e.g., heart, lung, pancreas).
* Organ transplant recipients or candidates.
* Hypersensitivity to interferon or excipients.
* Concurrent participation in other HBV-related interventional trials.
* Other conditions deemed unsuitable by investigators (e.g., non-compliance risk).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 30 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-05-31 (Estimated)

PRIMARY OUTCOMES:
HBV DNA and HBsAg undetectable with/without anti-HBs | week 72
  Proportion of patients achieving HBV DNA below the lower limit of quantification (LLOQ; <20 IU/mL), HBsAg undetectable (<0.05 IU/mL) (with or without anti-HBs seroconversion), and normal liver biochemical indices at Week 72.

SECONDARY OUTCOMES:
HBV DNA and HBsAg undetectable with/without anti-HBs during the study | Weeks 24, 48, and 96
  Proportion of patients achieving HBV DNA <20 IU/mL, HBsAg <0.05 IU/mL (with or without anti-HBs), and normal liver biochemistry at Weeks 24, 48, and 96.
HBV DNA and HBsAg undetectable during the study | Weeks 24, 48, 72, and 96
  Proportion of patients achieving HBsAg <0.05 IU/mL and HBV DNA <20 IU/mL at Weeks 24, 48, 72, and 96.
HBsAg level | Weeks 24, 48, 72, and 96
  HBsAg levels in each group at Weeks 24, 48, 72, and 96
HBsAg decline from baseline | Weeks 24, 48, 72, and 96
  Magnitude of HBsAg decline from baseline in each group at Weeks 24, 48, 72, and 96
HBsAg seroclearance | Weeks 24, 48, 72, and 96
  HBsAg seroclearance rate (HBsAg <0.05 IU/mL) in each group at Weeks 24, 48, 72, and 96
HBsAg seroconversion | Weeks 24, 48, 72, and 96
  HBsAg seroconversion rate (anti-HBs ≥10 mIU/mL) in each group at Weeks 24, 48, 72, and 96
HBeAg seroclearance | Weeks 24, 48, 72, and 96
  HBeAg seroclearance rate in baseline HBeAg-positive patients at Weeks 24, 48, 72, and 96
HBeAg seroconversion | Weeks 24, 48, 72, and 96
  HBeAg seroconversion rate (anti-HBe positivity) in baseline HBeAg-positive patients at Weeks 24, 48, 72, and 96
HBV DNA level | Weeks 24, 48, 72, and 96
  HBV DNA levels in each group at Weeks 24, 48, 72, and 96
HBV DNA decline from baseline | Weeks 24, 48, 72, and 96
  Magnitude of HBV DNA decline from baseline in each group at Weeks 24, 48, 72, and 96
HBV DNA undetectabe | Weeks 24, 48, 72, and 96
  HBV DNA undetectability rate (<20 IU/mL) in baseline HBV DNA-positive patients at Weeks 24, 48, 72, and 96
ALT levels | Weeks 24, 48, 72, and 96
  ALT levels in each group at Weeks 24, 48, 72, and 96
ALT normalization | Weeks 24, 48, 72, and 96
  ALT normalization rate (≤upper limit of normal [ULN]) in each group at Weeks 24, 48, 72, and 96
ALT levels from baseline | Weeks 24, 48, 72, and 96
  Change in ALT levels from baseline in each group at Weeks 24, 48, 72, and 96
saftey | Weeks 24, 48, 72, and 96
  Incidence of adverse events (AEs), serious adverse events (SAEs), and adverse drug reactions (ADRs) during the study, including findings from Physical examinations, Laboratory tests, Hematology, Urinalysis, Blood biochemistry, Coagulation profile

OTHER OUTCOMES:
HBV RNA | Weeks 24, 48, 72, and 96
  HBV pregenomic RNA (pgRNA) levels in each group at Weeks 24, 48, 72, and 96.
HBcrAg | Weeks 24, 48, 72, and 96
  HBV core-related antigen (HBcrAg) levels in each group at Weeks 24, 48, 72, and 96
HBsAg-specific T-cell and B-cell | during the study
  Longitudinal changes in HBsAg-specific T-cell and B-cell responses during the study
HBV quasispecies variations | Weeks 24, 48, 72, and 96
  Characterize HBV quasispecies variations
proteomic profiles | Weeks 24, 48, 72, and 96
  Assess longitudinal changes in proteomic profiles during the study
baseline GWAS | baseline
  Analyze baseline genomic characteristics and GWAS (Genome-Wide Association Study) data of patients

CONTACTS AND LOCATIONS:
Overall Officials: Wenghong Zhang, MD, Principal Investigator — Huashan Hospital; Jiming Zhang, MD, Principal Investigator — Huashan Hospital; Yuxian Huang, MD, Principal Investigator — Huashan Hospital; Feng Sun, MD, Study Chair — Huashan Hospital; Chao Qiu, Principal Investigator — Huashan Hospital; Chen Chen, MD, Study Director — Huashan Hospital; Qiran Zhang, MD, Study Director — Huashan Hospital
Locations (1):
- Huashan Hospita, Shanghai, China, China

REFERENCES:
- [Background] Ning Q, Han M, Sun Y, Jiang J, Tan D, Hou J, Tang H, Sheng J, Zhao M. Switching from entecavir to PegIFN alfa-2a in patients with HBeAg-positive chronic hepatitis B: a randomised open-label trial (OSST trial). J Hepatol. 2014 Oct;61(4):777-84. doi: 10.1016/j.jhep.2014.05.044. Epub 2014 Jun 7. PMID 24915612
- [Background] Yuen MF, Lim YS, Yoon KT, Lim TH, Heo J, Tangkijvanich P, Tak WY, Thanawala V, Cloutier D, Mao S, Arizpe A, Cathcart AL, Gupta SV, Hwang C, Gane E. VIR-2218 (elebsiran) plus pegylated interferon-alfa-2a in participants with chronic hepatitis B virus infection: a phase 2 study. Lancet Gastroenterol Hepatol. 2024 Dec;9(12):1121-1132. doi: 10.1016/S2468-1253(24)00237-1. Epub 2024 Oct 8. PMID 39389081
- [Background] Mak LY, Wooddell CI, Lenz O, Schluep T, Hamilton J, Davis HL, Mao X, Seto WK, Biermer M, Yuen MF. Long-term hepatitis B surface antigen response after finite treatment of ARC-520 or JNJ-3989. Gut. 2025 Feb 6;74(3):440-450. doi: 10.1136/gutjnl-2024-333026. PMID 39266050
- [Background] Buti M, Heo J, Tanaka Y, Andreone P, Atsukawa M, Cabezas J, Chak E, Coffin CS, Fujiwara K, Gankina N, Gordon SC, Janczewska E, Komori A, Lampertico P, McPherson S, Morozov V, Plesniak R, Poulin S, Ryan P, Sagalova O, Sheng G, Voloshina N, Xie Q, Yim HJ, Dixon S, Paff M, Felton L, Lee M, Greene T, Lim J, Lakshminarayanan D, McGonagle G, Plein H, Youssef AS, Elston R, Kendrick S, Theodore D. Sequential Peg-IFN after bepirovirsen may reduce post-treatment relapse in chronic hepatitis B. J Hepatol. 2025 Feb;82(2):222-234. doi: 10.1016/j.jhep.2024.08.010. Epub 2024 Aug 29. PMID 39214467
- [Background] Yuen MF, Lim SG, Plesniak R, Tsuji K, Janssen HLA, Pojoga C, Gadano A, Popescu CP, Stepanova T, Asselah T, Diaconescu G, Yim HJ, Heo J, Janczewska E, Wong A, Idriz N, Imamura M, Rizzardini G, Takaguchi K, Andreone P, Arbune M, Hou J, Park SJ, Vata A, Cremer J, Elston R, Lukic T, Quinn G, Maynard L, Kendrick S, Plein H, Campbell F, Paff M, Theodore D; B-Clear Study Group. Efficacy and Safety of Bepirovirsen in Chronic Hepatitis B Infection. N Engl J Med. 2022 Nov 24;387(21):1957-1968. doi: 10.1056/NEJMoa2210027. Epub 2022 Nov 8. PMID 36346079